CLINICAL TRIAL: NCT00883389
Title: Safe Kidney Care Med-Alert Bracelet/Keytag
Brief Title: Med-alert Bracelet in Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Jeffrey Fink, PI, University of Maryland, Baltimore
Other Study IDs: HP-00041163
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Results first posted 2012-08-21 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Chronic Kidney Disease
Keywords: patient safety; chronic kidney disease; med-alert
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Emergency Medical Tags

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Safe Kidney Care: Patients with Chronic Kidney Disease (eGFR < 60 ml/min/1.732)and not expected to need dialysis within 6 months of enrollment
  Interventions: Device: Medical Alert Bracelet

INTERVENTIONS:
Device: Medical Alert Bracelet — Medical Alert Bracelet alerting health care providers to consider the patient's chronic kidney disease condition when planning care. It also provides a link to a website about safe kidney care (safekidneycare.org)
  Other Names: Safe Kidney Care

SUMMARY:
This is a pilot observational study to evaluate subjects with chronic kidney disease acceptance of an alert device linked to an informational website intended to increase recognition of chronic kidney disease, and to guide patients and providers to the safe delivery of care required for this disease. Primary device was a bracelet with the alternative of a key fob with same information supplied when requested. Patients usage of the device was evaluated by survey with Likert scale as to whether the device is 0 = not useful, 1 = somewhat useful, 2 = extremely useful

DETAILED DESCRIPTION:
No need for more extensive description

ELIGIBILITY:
Inclusion Criteria:

* Persons with chronic kidney disease defined as estimated glomerular filtration rate of < 60 ml/min/1.73m2.

Exclusion Criteria:

* Persons expected to be on dialysis within 6 months.
* Less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic kidney disease and impaired kidney function
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2008-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey C Fink, MD MS, Principal Investigator — University of Maryland, College Park

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Medical records of renal patients screened for eligibility upon arrival of their clinic appointment. Patients meeting study criteria approached at the end of their appointment regarding their interest in participating
Pre-assignment Details: All recruited participants assigned to receive intervention (medical alert accessory)
Groups:
- Med-alert Bracelet Pilot Group: All participants assigned to the medical alert accessory group. There is no placebo
Period: Overall Study
Arm/Group | Med-alert Bracelet Pilot Group
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Med-alert Bracelet Pilot Group
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Qualitative Survey Assessmentof Perceived Usefulness of the Med-alert Device.
Description: Qualitative questionnaire with primary assessment: "How useful do you think the Med-alert device will be for future healthcare". Response recorded based on a Likert scale with response of 0 = not useful, 1 = somewhat useful, 2 = extremely useful
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: Likert scale
Groups:
- Med-alert Pilot Group: Participants in pilot study assigned a med-alert device of bracelet or necklace
Arm/Group | Med-alert Pilot Group
Number analyzed (Participants) | 24
Likert scale | 1 [1 to 2]

ADVERSE EVENTS:
Time Frame: 3 months
Description: Serious adverse events were collected if reported but not anticipated given the low risk of the medical alert device. Individuals at risk for such events were all those enrolled and were assessed in all this surveyed at 3 month time interval. None were reported.
Arm/Group | Med-alert Bracelet Pilot Group
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No